CLINICAL TRIAL: NCT05866731
Title: The Heart Rhythm Twins Study -- A Pilot Study in Identical and Fraternal Twins
Brief Title: The Heart Rhythm Twins Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 21-35126
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Premature Atrial Complex; Premature Ventricular Contraction
Keywords: twin
MeSH Terms: conditions — Atrial Premature Complexes; Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Identical twins: 60 identical twins (30 sets) will be enrolled. Participants will answer 15-20 minutes of questionnaires on demographics, lifestyle, medical history, and family history over Zoom or the phone with a study coordinator. Participants will then be mailed an iRhythm Zio XT heart rhythm monitor, or EKG, to apply and wear for a maximum of 2 weeks, as well as a DNA Genotek saliva collection kit to collect a small saliva sample. Participants will return the monitor and saliva sample to the study team, and will be reimbursed upon return. The study team is also requesting photo validation to verify twin status.
- Same-sex fraternal twins: 60 same-sex fraternal twins (30 sets) will be enrolled. Participants will answer 15-20 minutes of questionnaires on demographics, lifestyle, medical history, and family history over Zoom or the phone with a study coordinator. Participants will then be mailed an iRhythm Zio XT heart rhythm monitor, or EKG, to apply and wear for a maximum of 2 weeks, as well as a DNA Genotek saliva collection kit to collect a small saliva sample. Participants will return the monitor and saliva sample to the study team, and will be reimbursed upon return. The study team is also requesting photo validation to verify twin status.

SUMMARY:
Premature atrial contractions (PACs) and premature ventricular contractions (PVCs) are observed in the majority of individuals monitored for more than a few hours. Although the clinical course of PACs and PVCs is usually benign, it has been described that high PAC or PVC frequency causes various comorbidities and worsens outcomes in different patient groups. For example, PACs can initiate episodes of atrial fibrillation, and PAC count is highly specific in predicting diagnosis of incident atrial fibrillation. Increasing PVC frequencies are an important predictor of incident heart failure.

While conventional wisdom dictates that common environmental exposures determine PAC and PVC frequencies, this has not born out in rigorous studies. Whether PAC and PVC frequencies may have genetic underpinnings remains unknown.

Comparisons between identical twins and fraternal twins can provide estimates of heritability. Fraternal twins are an ideal control because, like identical twins, they share a womb, have the same birthday, and their environment while growing up are as similar as between identical twins. However, while identical twins share approximately 100% of the same inherited DNA, fraternal twins share, on average, about 50%. By monitoring identical and fraternal twins with portable electrocardiograms (ECGs), we will be able to count the PACs and PVCs over a consecutive timespan to describe the familial aggregation of these complexes. This, to our knowledge, would be the first study to compare PAC and PVC frequencies in identical and same-sex fraternal twins, providing the first assessment of how genetical inheritance may influence cardiac ectopy burdens.

ELIGIBILITY:
Inclusion Criteria:

* Identical or same-sex fraternal sets of twins
* English-speaking

Exclusion Criteria:

* Pregnancy
* Current anti-arrhythmic medication use (including beta blockers)
* Diagnosis of congenital heart disease
* Diagnosis of persistent or permanent atrial fibrillation
* Prior cardiac ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Same-sex sets of twins from anywhere in the world can enroll, as all study procedures can be done remotely. Both twins must enroll to participate.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of premature atrial contractions (PACs) | Maximum of 2 weeks
  This will be measured using a wearable EKG monitor.
Frequency of premature ventricular contractions (PVCs) | Maximum of 2 weeks
  This will be measured using a wearable EKG monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Marcus, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No